CLINICAL TRIAL: NCT01022424
Title: A Long-term Administration Study of OPC-41061 in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) (2) [Extension of Study 156-05-002]
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-09-003; JapicCTI-090948 (Other: JAPIC)
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD; Tolvaptan; OPC-41061
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-41061 (Experimental): Repeated oral administration at doses of 15 mg twice daily (morning and evening)
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061 — Repeated oral administration at doses of 15 mg twice daily (morning and evening)

SUMMARY:
ADPKD patients who were enrolled in Study 156-05-002 will receive repeated oral administration of OPC-41061 at doses of 15 mg twice daily (morning and evening). Administration will be continued until the time of manufacturing and distribution approval of OPC-41061 for ADPKD in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed 3-year repeated administrations and the follow-up observation or those who were withdrawn from the study due to reasons other than occurrence of adverse events (based on the judgment of either the subject or the investigator/subinvestigator) in the preceding study (156-05-002)
* Patients in whom adverse events occurring in study 156-05-002 were resolved or became stable and do not require further follow-up.

Exclusion Criteria:

* Patients with eGFR of less than 15 mL/min/1.73 m2
* Patients with any of the following complications:

  * Uncontrolled hypertension
  * Serious cardiovascular disease (eg. heart failure) or hepatic disease (eg. cirrhosis)
* Patients with any of the following complications or history thereof:

  * Clinically significant drug allergies (anaphylaxis) or hypersensitivity (especially, hypersensitivity to benzazepine derivatives or suspected hypersensitivity
  * Inability to personally give consent due to a mental illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanto Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-41061: Repeated oral administration at doses of 15 mg twice daily (morning and evening) until approval of the revised protocol (Edition 4.0) by the IRB of each trial site.
  Repeated oral administration at one of three split dose-regimens 45mg/15mg, 60mg/30mg or 90mg/30mg twice daily (morning and evening) following approval of the revised protocol.
Period: Overall Study
Arm/Group | OPC-41061
Started | 13
Completed | 9
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — eGFR under the withdrawal criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | OPC-41061
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  Japan | 13

OUTCOME MEASURES:

1. Primary Outcome: Total Kidney Volume
Description: Individual subject data on the volumes of the total kidney volume (sum of the volumes of the left and right kidneys) measured by magnetic resonance imaging or computed tomography during trial period.
  Repeated oral administration at doses of 15 mg twice daily (morning and evening) until approval of the revised protocol (Edition 4.0) by the IRB of each trial site.
  Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, Week 48, 96, 144, and 192
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Baseline; Week 48; Week 96; Week 144; Week 192: Repeated oral administration at doses of 15 mg twice daily (morning and evening) until approval of the revised protocol (Edition 4.0) by the IRB of each trial site.
  Repeated oral administration at one of three split dose-regimens 45mg/15mg, 60mg/30mg or 90mg/30mg twice daily (morning and evening) following approval of the revised protocol.
Arm/Group | Baseline | Week 48 | Week 96 | Week 144 | Week 192
Number analyzed (Participants) | 13 | 12 | 12 | 11 | 10
mL | 1428 [789 to 4774] | 1675 [786 to 4457] | 1728 [791 to 4193] | 1775 [818 to 4125] | 1901 [837 to 3669]

2. Primary Outcome: Renal Function Test (eGFR)
Description: Individual subject data on eGFR (estimated glomerular filtration rate calculated by Japanese eGFR equation) during trial period.
  Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, Week 48, 96, 144, and 192
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73 m2
Arm/Group | Baseline | Week 48 | Week 96 | Week 144 | Week 192
Number analyzed (Participants) | 13 | 12 | 12 | 11 | 10
mL/min/1.73 m2 | 63.0 [31.0 to 93.0] | 60.0 [23.0 to 92.0] | 54.0 [22.0 to 113.0] | 50.5 [15.0 to 63.0] | 51.0 [16.0 to 64.0]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 years
Arm/Group | OPC-41061
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 (N=13)
Retinal vein occlusion (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Hepatic cyst infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Alcoholism (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 (N=13)
Anaemia (Blood and lymphatic system disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Angle closure glaucoma (Eye disorders) | 1
Asthenopia (Eye disorders) | 1
Cataract (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Meibomianitis (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Eyelids pruritus (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 2
Hyperchlorhydria (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 3
Thirst (General disorders) | 6
Biliary cirrhosis primary (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Acute tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 8
Periodontitis (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Hepatic cyst infection (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood antidiuretic hormone increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood osmolarity increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Electrocardiogram T wave inversion (Investigations) | 1
Haematocrit increased (Investigations) | 1
Haemoglobin increased (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Red blood cell count increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Cystatin C increased (Investigations) | 1
Urinary casts present (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hyperaesthesia (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Eating disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 4
Polyuria (Renal and urinary disorders) | 3
Renal cyst haemorrhage (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Endometriosis (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Chloasma (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Urticaria cholinergic (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No